CLINICAL TRIAL: NCT03978520
Title: A Phase 2 Study to Investigate the Safety and Efficacy of Elsubrutinib and Upadacitinib Given Alone or in Combination (ABBV-599 Combination) in Subjects With Moderately to Severely Active Systemic Lupus Erythematosus
Brief Title: A Study to Investigate the Safety and Efficacy of Elsubrutinib and Upadacitinib Given Alone or in Combination in Participants With Moderately to Severely Active Systemic Lupus Erythematosus (SLE)
Acronym: SLEek
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M19-130; 2019-000638-20 (EudraCT Number)
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-06

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: Systemic Lupus Erythematosus (SLE); ABBV-105; Upadacitinib; ABBV-599; Elsubrutinib
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Elsubrutinib placebo/upadacitinib placebo (Placebo Comparator): Placebo capsule for elsubrutinib once a day by mouth for up to 48 weeks; placebo film-coated tablet for upadacitinib once a day by mouth for up to 48 weeks
  Interventions: Drug: Placebo for elsubrutinib; Drug: Placebo for upadacitinib
- ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) (Experimental): 60 mg elsubrutinib capsule once a day by mouth for up to 48 weeks; 30 mg upadacitinib film-coated tablet once a day by mouth for up to 48 weeks
  Interventions: Drug: Elsubrutinib; Drug: Upadacitinib
- Elsubrutinib placebo/upadacitinib 30 mg (Experimental): Placebo capsule for elsubrutinib once a day by mouth for up to 48 weeks; 30 mg upadacitinib film-coated tablet once a day by mouth for up to 48 weeks
  Interventions: Drug: Placebo for elsubrutinib; Drug: Upadacitinib
- ABBV-599 Low Dose (Elsubrutinib 60 mg/upadacitinib 15 mg) (Experimental): 60 mg elsubrutinib capsule once a day by mouth for up to 24 weeks; 15 mg upadacitinib film-coated tablet once a day by mouth for up to 24 weeks
  Interventions: Drug: Elsubrutinib; Drug: Upadacitinib
- Elsubrutinib 60 mg/upadacitinib placebo (Experimental): 60 mg elsubrutinib capsule once a day by mouth for up to 24 weeks; placebo film-coated tablet for upadacitinib once a day by mouth for up to 24 weeks
  Interventions: Drug: Elsubrutinib; Drug: Placebo for upadacitinib

INTERVENTIONS:
Drug: Elsubrutinib — Capsule; Oral
  Other Names: ABBV-105
  Arms: ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg); ABBV-599 Low Dose (Elsubrutinib 60 mg/upadacitinib 15 mg); Elsubrutinib 60 mg/upadacitinib placebo
Drug: Placebo for elsubrutinib — Capsule; Oral
  Arms: Elsubrutinib placebo/upadacitinib 30 mg; Elsubrutinib placebo/upadacitinib placebo
Drug: Upadacitinib — Film-coated tablet; Oral
  Other Names: RINVOQ
  Arms: ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg); ABBV-599 Low Dose (Elsubrutinib 60 mg/upadacitinib 15 mg); Elsubrutinib placebo/upadacitinib 30 mg
Drug: Placebo for upadacitinib — Film-coated tablet; Oral
  Arms: Elsubrutinib 60 mg/upadacitinib placebo; Elsubrutinib placebo/upadacitinib placebo

SUMMARY:
The main objective of this study was to evaluate the safety and efficacy of elsubrutinib, upadacitinib (UPA), and ABBV-599 (elsubrutinib/upadacitinib) High Dose and Low Dose combinations vs placebo for the treatment of signs and symptoms of Systemic Lupus Erythematosus (SLE) in participants with moderately to severely active SLE and to define doses for further development.

ELIGIBILITY:
Inclusion Criteria:

* Participant has clinical diagnosis of Systemic Lupus Erythematosus (SLE) at least 24 weeks prior to Screening, meeting at least 4 of the 11 revised Criteria for Classification of SLE according to the 1997 Update of the 1982 American College of Rheumatology (ACR) OR meeting at least 4 of the 2012 SLICC classification criteria, including at least 1 clinical criterion and 1 immunologic criterion.
* At Screening, must have at least one of the following:

  * antinuclear antibody (ANA)+ (titer ≥ 1:80)
  * anti-dsDNA+
  * anti-Smith+
* SLEDAI-2K (SLE Disease Activity Index) ≥ 6 despite background therapy as reported and independently adjudicated (clinical score ≥ 4, excluding lupus headache and/or organic brain syndrome) at Screening:

  * If 4 points of the required entry points are for arthritis, there must also be a minimum of 3 tender and 3 swollen joints.
  * If participant has rash and Principal Investigator (PI) considers it to be attributable to SLE, participant must consent to skin photograph collection for adjudication.
  * Score must be re-confirmed at the Baseline visit.
* Physician's Global Assessment (PhGA) ≥ 1 during screening period.
* Must be on background treatment, stable for 30 days prior to Baseline and throughout the study with antimalarial(s), prednisone (or prednisone equivalent) (≤ 20 mg), azathioprine (≤ 150 mg), mycophenolate (<2 g), leflunomide (≤ 20 mg), cyclosporine, tacrolimus, and/or methotrexate (MTX) (≤ 20 mg).

  * No combinations of the above with immunomodulators other than prednisone (or equivalents) and antimalarials.

Exclusion Criteria:

- Participant using intravenous (IV) or intramuscular (IM) corticosteroids greater than or equal to a 40 mg prednisone-equivalent bolus within 30 days of planned randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (160):
- United States (47):
  - Arizona Arthritis & Rheumatology Research, PLLC /ID# 214522, Mesa, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 211329, Phoenix, Arizona
  - AZ Arthritis and Rheumotology Research, PLLC /ID# 214267, Phoenix, Arizona
  - Arthritis and Rheumatism Associates /ID# 211411, Jonesboro, Arkansas
  - Wallace Rheumatic Studies Center, LLC /ID# 211600, Beverly Hills, California
  - Arthritis & Osteo Medical Ctr /ID# 228235, La Palma, California
  - Valerius Medical Group & Research Center /ID# 211599, Los Alamitos, California
  - East Bay Rheumatology Medical /ID# 211638, San Leandro, California
  - The Lundquist Institute at Harbor-UCLA Medical Center /ID# 213402, Torrance, California
  - Medvin Clinical Research /ID# 211996, Tujunga, California
  - Inland Rheum Clin Trials Inc. /ID# 213617, Upland, California
  - University of Colorado Hospital /ID# 211314, Aurora, Colorado
  - Yale University /ID# 212824, New Haven, Connecticut
  - Medstar Health Research Institute /ID# 213335, Washington D.C., District of Columbia
  - Arthritis & Rheumatic Disease Specialties /ID# 214052, Aventura, Florida
  - LeJenue Research Associates /ID# 212327, Miami, Florida
  - Ctr Arthritis & Rheumatic Dise /ID# 212326, Miami, Florida
  - Millennium Research /ID# 219099, Ormond Beach, Florida
  - IRIS Research and Development, LLC /ID# 213053, Plantation, Florida
  - West Broward Rheumatology Associates /ID# 211881, Tamarac, Florida
  - BayCare Medical Group, Inc. /ID# 218818, Tampa, Florida
  - Affinity Clinical Research /ID# 211496, Oak Brook, Illinois
  - Deerbrook Medical Associates /ID# 212251, Vernon Hills, Illinois
  - Qualmedica Research, LLC /ID# 214765, Evansville, Indiana
  - University of Iowa Hospitals and Clinics /ID# 215246, Iowa City, Iowa
  - The Center for Rheumatology and Bone Research /ID# 211610, Wheaton, Maryland
  - Beth Israel Deaconess Medical Center /ID# 212321, Boston, Massachusetts
  - Henry Ford Health System /ID# 211676, Detroit, Michigan
  - June DO, PC /ID# 211674, Lansing, Michigan
  - West County Rheumatology /ID# 225051, St Louis, Missouri
  - NYU Langone Ambulatory Care Brooklyn Heights /ID# 211548, Brooklyn, New York
  - NYU Langone Orthopedic Center /ID# 213620, New York, New York
  - Ohio State University - Wexner Medical Center /ID# 211636, Columbus, Ohio
  - STAT Research, Inc. /ID# 211404, Vandalia, Ohio
  - Premier Rheumatology of Oklahoma /ID# 213850, Tulsa, Oklahoma
  - Allegheny Health Network Research Institute /ID# 211607, Pittsburgh, Pennsylvania
  - Univ TN Health Sciences Ctr /ID# 212177, Memphis, Tennessee
  - Dr. Ramesh Gupta /ID# 213381, Memphis, Tennessee
  - Tekton Research, Inc. /ID# 211521, Austin, Texas
  - Tekton Research, Inc. /ID# 214182, Austin, Texas
  - Trinity Universal Research Associates - Carrollton /ID# 211527, Carrollton, Texas
  - Accurate Clinical Management /ID# 213571, Houston, Texas
  - West Texas Clinical Research /ID# 211529, Lubbock, Texas
  - SW Rheumatology Res. LLC /ID# 211520, Mesquite, Texas
  - Carilion Clinic /ID# 213500, Roanoke, Virginia
  - Virginia Mason Medical Center /ID# 211457, Seattle, Washington
  - Rheumatology and Pulmonary Clinic /ID# 211398, Beckley, West Virginia
- Argentina (9):
  - Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich /ID# 221685, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Interzonal General de Agudos General Jose de San Martin /ID# 211679, La Plata, Buenos Aires
  - CER Instituto Medico /ID# 222757, Quilmes, Buenos Aires
  - Aprillus Asistencia e Investigacion /ID# 211630, Ciudad Autonoma de Buenos Aire, Ciuadad Autonoma de Buenos Aires
  - Centro de Enfermedades del Hígado y Aparato Digestivo /ID# 211634, Rosario, Santa Fe Province
  - Instituto CAICI S.R.L /ID# 211633, Rosario, Santa Fe Province
  - Centro de Investigaciones Medicas Tucuman /ID# 212714, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clinicas Tucuman /ID# 211942, San Miguel de Tucumán, Tucumán Province
  - Hospital Cordoba /ID# 212200, Córdoba
- Australia (9):
  - Emeritus Research Sydney /ID# 222983, Botany, New South Wales
  - Royal North Shore Hospital /ID# 222982, St Leonards, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 212667, Herston, Queensland
  - Rheumatology Research Unit Sunshine Coast /ID# 211902, Maroochydore, Queensland
  - Griffith University /ID# 223543, Southport, Queensland
  - The Queen Elizabeth Hospital /ID# 211901, Woodville South, South Australia
  - Emeritus Research /ID# 211903, Camberwell, Victoria
  - Monash Medical Centre /ID# 212313, Clayton, Victoria
  - St Vincent's Hospital Melbourne /ID# 212311, Fitzroy Melbourne, Victoria
- Bulgaria (3):
  - UMHAT Kaspela EOOD /ID# 223141, Plovdiv
  - UMHAT Sveti Ivan Rilski /ID# 223139, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 223140, Sofia
- Canada (4):
  - Hamilton Health Sciences - McMaster University Medical Centre /ID# 212662, Hamilton, Ontario
  - St. Josephs Health Care Centre /ID# 212331, London, Ontario
  - Toronto Western Hospital /ID# 213336, Toronto, Ontario
  - Diex Recherche Sherbrooke Inc. /ID# 217734, Sherbrooke, Quebec
- China (8):
  - Anhui Provincial Hospital /ID# 211812, Hefei, Anhui
  - Peking Union Medical College Hospital /ID# 211614, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital /ID# 211811, Guangzhou, Guangdong
  - Xiangya Hospital Central South University /ID# 212919, Changsha, Hunan
  - Jiangsu Province Hospital /ID# 211818, Nanjing, Jiangsu
  - Huashan Hospital, Fudan University /ID# 213976, Shanghai, Shanghai Municipality
  - Shanghai Changhai Hospital /ID# 211819, Shanghai, Shanghai Municipality
  - People's Hospital of Xinjiang /ID# 211821, Ürümqi
- Colombia (5):
  - Centro Integral de Reumatologia del Caribe Circaribe SAS /ID# 211894, Barranquilla, Atlántico
  - Centro de Investigacion en Reumatologia y Especialidades Medicas- CIREEM SAS /ID# 211895, Bogota, Cundinamarca
  - Preventive Care Sas /Id# 211896, Chía, Cundinamarca
  - Healthy Medical Center SAS /ID# 211899, Zipaquirá, Cundinamarca
  - Clinica Universitaria Bolivari /ID# 211897, Medellín
- France (5):
  - CHRU Lille - Hopital Claude Huriez /ID# 211829, Lille, Hauts-de-France
  - CHU Bordeaux - Hopital Pellegrin /ID# 211832, Bordeaux
  - AP-HP - Hôpital Bicêtre /ID# 211968, Le Kremlin-Bicêtre
  - Hopital Pitie Salpetriere /ID# 211831, Paris
  - CHU Strasbourg - Hopital Civil /ID# 211981, Strasbourg
- Germany (4):
  - Universitaetsklinikum Duesseldorf /ID# 212408, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 212674, Kiel, Schleswig-Holstein
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 211988, Berlin
  - Universitaetsklinikum Carl Gustav Carus an der TU Dresden /ID# 212770, Dresden
- Hungary (4):
  - Debreceni Egyetem Klinikai Kozpont /ID# 212042, Debrecen, Hajdú-Bihar
  - Vital Medical Center Orvosi es Fogaszati Kozpont /ID# 212796, Veszprém, Veszprém megye
  - Orszagos Reumatologiai es Fizioterapias Intezet /ID# 211827, Budapest
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaz /ID# 216971, Gyula
- Italy (4):
  - Azienda Ospedaliero-Universitaria di Ferrara-Arcispedale Sant Anna /ID# 211861, Cona, Ferrara
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 212195, Rome, Lazio
  - ASST Gaetano Pini/Presidio Ospedaliero Pini /ID# 215063, Milan
  - Azienda Ospedaliera Universitaria Friuli Centrale/Presidio Ospedaliero Universit /ID# 211858, Udine
- Japan (17):
  - Chukyo Hospital /ID# 222625, Nagoya, Aichi-ken
  - NHO Nagoya Medical Center /ID# 213974, Nagoya, Aichi-ken
  - Hamanomachi Hospital /ID# 213696, Fukuoka, Fukuoka
  - Hospital of the University of Occupational and Environmental Health, Japan /ID# 217548, Kitakyushu-shi, Fukuoka
  - Fukushima Medical University Hospital /ID# 213913, Fukushima, Fukushima
  - Hiroshima Red Cross Hospital & Atomic-bomb Survivors Hospital /ID# 213694, Hiroshima, Hiroshima
  - National Hospital Organization Asahikawa Medical Center /ID# 213846, Asahikawa-shi, Hokkaido
  - Tomakomai City Hospital /ID# 214234, Tomakomai-shi, Hokkaido
  - Kita-harima Medical Center /ID# 215474, Ono-shi, Hyōgo
  - EIRAKU Internal Medicine Clinic /ID# 215419, Kagoshima, Kagoshima-ken
  - Yokohama Rosai Hospital /ID# 213690, Yokohama, Kanagawa
  - Kumamoto Shinto General Hospital /ID# 215347, Kumamoto, Kumamoto
  - Tohoku University Hospital /ID# 213693, Sendai, Miyagi
  - Shinshu University Hospital /ID# 213853, Matsumoto-shi, Nagano
  - Nagano Red Cross Hospital /ID# 214572, Nagano, Nagano
  - Saitama Medical Center /ID# 213687, Kawagoe-shi, Saitama
  - Keio University Hospital /ID# 216347, Shinjuku-ku, Tokyo
- Mexico (7):
  - Morales Vargas Centro de Investigacion S.C. /ID# 212946, León, Guanajuato
  - Centro Integral en Reumatologia S.A de C.V /ID# 211876, Guadalajara, Jalisco
  - Centro de Estudios de Investigación Básica y Clínica, S.C. /ID# 212532, Guadalajara, Jalisco
  - RM Pharma Specialists S.A de C.V. /ID# 211879, Mexico City, Mexico City
  - CINTRE, Centro de Investigación y Tratamiento Reumatológico SC /ID# 211875, Mexico City, Mexico City
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí, SC /ID# 212737, San Luis Potosí City, San Luis Potosí
  - Medical Care & Research SA de CV /ID# 212682, Mérida, Yucatán
- Netherlands (3):
  - Vrije Universiteit Medisch Centrum /ID# 214424, Amsterdam
  - Leids Universitair Medisch Centrum /ID# 214413, Leiden
  - Universitair Medisch Centrum Utrecht /ID# 214415, Utrecht
- New Zealand (3):
  - Middlemore Clinical Trials /ID# 213504, Papatoetoe, Auckland
  - North Shore Hospital /ID# 213506, Takapuna, Auckland
  - Waikato Hospital /ID# 213505, Hamilton, Waikato Region
- Poland (4):
  - Ortopedyczno-Rehabilitacyjny Szpital Kliniczny im. Wiktora Degi /ID# 212483, Poznan, Greater Poland Voivodeship
  - Centrum Nowoczesnych Terapii Dobry Lekarz Sp. z o.o. /ID# 212146, Krakow, Lesser Poland Voivodeship
  - WroMedica I. Bielicka, A. Strzalkowska s.c. /ID# 212482, Wroclaw, Lower Silesian Voivodeship
  - Centrum Medyczne Pratia Warszawa /ID# 218176, Warsaw, Masovian Voivodeship
- Puerto Rico (2):
  - GCM Medical Group PSC /ID# 211251, San Juan
  - Mindful Medical Research /ID# 213384, San Juan
- South Korea (5):
  - Ajou University Hospital /ID# 211692, Suwon, Gyeonggido
  - KonKuk University Medical Center /ID# 213410, Seoul, Seoul Teugbyeolsi
  - Chonnam National University Hospital /ID# 211695, Gwangju
  - Inha University Hospital /ID# 211691, Incheon
  - Seoul National University Hospital /ID# 211740, Seoul
- Spain (8):
  - HUA - Txagorritxu /ID# 212520, Vitoria-Gasteiz, Alava
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 212145, Sabadell, Barcelona
  - Hospital Universitario Basurto /ID# 212722, Bilbao, Vizcaya
  - Hospital Universitario de Galdakao /ID# 212803, Galdakao, Vizcaya
  - Hospital Universitario A Coruna - CHUAC /ID# 211719, A Coruña
  - Hospital Universitario 12 de Octubre /ID# 211757, Madrid
  - Hospital Universitario Virgen de Valme /ID# 212721, Seville
  - Hospital Universitario y Politecnico La Fe /ID# 211720, Valencia
- Taiwan (6):
  - China Medical University Hospital /ID# 212179, Taichung
  - Taichung Veterans General Hospital /ID# 211957, Taichung
  - National Taiwan University Hospital /ID# 211752, Taipei
  - Taipei Medical University Hospital /ID# 221600, Taipei
  - Taipei Veterans General Hosp /ID# 212216, Taipei
  - Linkou Chang Gung Memorial Hospital /ID# 211751, Taoyuan
- United Kingdom (3):
  - Guys and St Thomas NHS Foundation Trust /ID# 211931, London, London, City of
  - Cambridge University Hospitals NHS Foundation Trust /ID# 213189, Cambridge
  - Manchester University NHS Foundation Trust /ID# 211838, Manchester

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Full Analysis Set: all randomized participants who received at least 1 dose of study drug
Period: Overall Study
Arm/Group | Elsubrutinib Placebo/Upadacitinib Placebo | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) | Elsubrutinib Placebo/Upadacitinib 30 mg | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) | Elsubrutinib 60 mg/Upadacitinib Placebo
Started | 75 | 68 | 62 | 69 | 67
Completed | 52 | 52 | 51 | 24 | 29
Not Completed | 23 | 16 | 11 | 45 | 38
Not completed — Adverse Event | 2 | 5 | 3 | 5 | 6
Not completed — Withdrawal by Subject | 10 | 4 | 5 | 6 | 5
Not completed — Lost to Follow-up | 2 | 2 | 2 | 0 | 1
Not completed — COVID-19 infection | 0 | 1 | 0 | 0 | 0
Not completed — Other, not specified | 9 | 4 | 1 | 1 | 2
Not completed — Sponsor decision based on interim analysis data review | 0 | 0 | 0 | 33 | 24

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Elsubrutinib Placebo/Upadacitinib Placebo | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) | Elsubrutinib Placebo/Upadacitinib 30 mg | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) | Elsubrutinib 60 mg/Upadacitinib Placebo | Total
Number analyzed (Participants) | 75 | 68 | 62 | 69 | 67 | 341
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (12.05) | 42.7 (11.27) | 42.5 (11.89) | 41.4 (11.85) | 42.0 (11.84) | 42.1 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 62 | 57 | 63 | 62 | 319
  Male | 0 | 6 | 5 | 6 | 5 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 0 | 1 | 4 | 11
  Asian | 23 | 14 | 13 | 13 | 9 | 72
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 9 | 8 | 6 | 31
  White | 43 | 45 | 34 | 45 | 44 | 211
  More than one race | 2 | 2 | 6 | 2 | 4 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score [Mean (Standard Deviation); unit: units on a scale] — The SLEDAI-2K is a global SLE disease activity index that focuses on high-impact disease manifestations across 9 organ systems. It includes 24 clinical and laboratory variables with manifestations weighted by the affected organ system. Scores range from 0 to 105, with higher scores indicating more severe disease.
  units on a scale | 9.1 (3.88) | 8.9 (2.75) | 9.0 (2.75) | 8.8 (2.86) | 9.2 (3.18) | 9.0 (3.12)
Physician's Global Assessment (PhGA) score [Mean (Standard Deviation); unit: units on a scale] — Physician's assessment of patient's overall disease activity due to Systemic Lupus Erythematosus (SLE), as compared with all possible participants with SLE. The benchmarks of the visual analog scale are 0, 1, 2, and 3 on the line corresponding to no, mild, moderate, and severe SLE disease activity, respectively.
  units on a scale | 1.75 (0.440) | 1.80 (0.417) | 1.70 (0.438) | 1.77 (0.422) | 1.77 (0.392) | 1.76 (0.421)
Daily dose of corticosteroid [Mean (Standard Deviation); unit: mg/day] | 7.937 (7.1270) | 6.743 (6.3736) | 6.242 (6.0920) | 6.891 (6.1056) | 6.291 (6.1096) | 6.856 (6.3885)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving SLE Responder Index (SRI)-4 and Steroid Dose ≤ 10 mg Prednisone Equivalent Once a Day (QD) at Week 24
Description: SLE Responder Index (SRI)-4 is defined as follows with all criteria compared to Baseline:
  * ≥ 4-point reduction in Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score
  * No worsening of the overall condition (< 0.3 point increase in Physician's Global Assessment [PhGA])
  * No new British Isles Lupus Assessment Group (BILAG) A or more than 1 new BILAG B disease activity scores (i.e., no organ system changes from baseline B/C/D/E to A and no more than 1 organ system changes from baseline C/D/E to B). A letter score is assigned to each organ system with following indications: A = severe, B = moderate, C = mild, D = inactive with prior history, and E = inactive with no history.
Time Frame: Baseline, Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug; non-responder imputation incorporating multiple imputation to handle missing data due to COVID-19 (NRI-C). When 50% of planned participants had completed Week 24 or withdrawn from the study, the ABBV-599 Low Dose and elsubrutinib 60 mg treatment groups were terminated as these groups did not meet projected efficacy. Per protocol, terminated groups were removed from the efficacy analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elsubrutinib Placebo/Upadacitinib Placebo | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) | Elsubrutinib Placebo/Upadacitinib 30 mg
Number analyzed (Participants) | 75 | 68 | 62
percentage of participants | 37.3 [26.4 to 48.3] | 48.5 [36.7 to 60.4] | 54.8 [42.5 to 67.2]
Statistical Analysis 1: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg); ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs elsubrutinib placebo/upadacitinib placebo The difference between the groups was assessed using the Cochran-Mantel-Haenszel (CMH) test, stratified by baseline corticosteroid dose above 10 mg prednisone-equivalent (≤10 mg or > 10 mg), screening SLEDAI-2K (< 10 or ≥10), baseline interferon score (high or low or NA), baseline immunosuppressant (azathioprine, tacrolimus, cyclosporine, methotrexate [MTX], mycophenolate) (yes or no); Test type: Superiority; p = 0.081, Cochran-Mantel-Haenszel; Response Rate Difference = 12.8, 95% CI 2-sided [-1.6 to 27.1]
Statistical Analysis 2: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs Elsubrutinib Placebo/Upadacitinib 30 mg; Elsubrutinib placebo/upadacitinib 30 mg vs elsubrutinib placebo/upadacitinib placebo The difference between the groups was assessed using the Cochran-Mantel-Haenszel (CMH) test, stratified by baseline corticosteroid dose above 10 mg prednisone-equivalent (≤10 mg or > 10 mg), screening SLEDAI-2K (< 10 or ≥10), baseline interferon score (high or low or NA), baseline immunosuppressant (azathioprine, tacrolimus, cyclosporine, methotrexate [MTX], mycophenolate) (yes or no); Test type: Superiority; p = 0.028, Cochran-Mantel-Haenszel; Response Rate Difference = 16.9, 95% CI 2-sided [1.8 to 31.9]
Statistical Analysis 3: Comparison: ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) vs Elsubrutinib Placebo/Upadacitinib 30 mg; ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs elsubrutinib placebo/upadacitinib 30 mg The difference between the groups was assessed using the Cochran-Mantel-Haenszel (CMH) test, stratified by baseline corticosteroid dose above 10 mg prednisone-equivalent (≤10 mg or > 10 mg), screening SLEDAI-2K (< 10 or ≥10), baseline interferon score (high or low or NA), baseline immunosuppressant (azathioprine, tacrolimus, cyclosporine, methotrexate [MTX], mycophenolate) (yes or no); Test type: Superiority; p = 0.566, Cochran-Mantel-Haenszel; Response Rate Difference = -4.7, 95% CI 2-sided [-20.8 to 11.4]

2. Secondary Outcome: Percentage of Participants Achieving SLE Responder Index (SRI)-4 at Week 24
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elsubrutinib Placebo/Upadacitinib Placebo | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) | Elsubrutinib Placebo/Upadacitinib 30 mg
Number analyzed (Participants) | 75 | 68 | 62
percentage of participants | 38.7 [27.6 to 49.7] | 54.4 [42.6 to 66.2] | 56.5 [44.1 to 68.8]
Statistical Analysis 1: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.013, Cochran-Mantel-Haenszel; Response Rate Difference = 18.3, 95% CI 2-sided [3.9 to 32.6]
Statistical Analysis 2: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs Elsubrutinib Placebo/Upadacitinib 30 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.018, Cochran-Mantel-Haenszel; Response Rate Difference = 18.1, 95% CI 2-sided [3.0 to 33.2]
Statistical Analysis 3: Comparison: ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) vs Elsubrutinib Placebo/Upadacitinib 30 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.882, Cochran-Mantel-Haenszel; Response Rate Difference = -1.2, 95% CI 2-sided [-17.6 to 15.2]

3. Secondary Outcome: Percentage of Participants Achieving British Isles Lupus Assessment Group (BILAG) Based Combined Lupus Assessment (BICLA) Response at Week 24
Description: BICLA is a composite responder index. Achievement of BICLA response is defined as improvement in all initial A and B BILAG scores, with no more than one new BILAG B score without worsening of the overall condition (no worsening in Physician's Global Assessment [PhGA], < 0.3 point increase) and no worsening of the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elsubrutinib Placebo/Upadacitinib Placebo | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) | Elsubrutinib Placebo/Upadacitinib 30 mg
Number analyzed (Participants) | 75 | 68 | 62
percentage of participants | 42.7 [31.5 to 53.9] | 54.4 [42.6 to 66.2] | 58.1 [45.8 to 70.3]
Statistical Analysis 1: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.049, Cochran-Mantel-Haenszel; Response Rate Difference = 14.7, 95% CI 2-sided [0.0 to 29.4]
Statistical Analysis 2: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs Elsubrutinib Placebo/Upadacitinib 30 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.091, Cochran-Mantel-Haenszel; Response Rate Difference = 13.9, 95% CI 2-sided [-2.2 to 30.1]
Statistical Analysis 3: Comparison: ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) vs Elsubrutinib Placebo/Upadacitinib 30 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.447, Cochran-Mantel-Haenszel; Response Rate Difference = -6.3, 95% CI 2-sided [-22.5 to 9.9]

4. Secondary Outcome: Percentage of Participants Achieving Lupus Low Disease Activity State (LLDAS) at Week 24
Description: LLDAS is a state of low disease activity based on Systemic Lupus Erythematosus Disease Activity Index 2000 score (SLEDAI-2K score ≤4 excluding SLEDAI-2K activity in major organ systems), absence of SLE disease activity in major organ systems and new disease activity, Physician's Global Assessment (PhGA ≤1), and concomitant medication usage (steroid dose ≤7.5 mg QD and toleration of immunosuppressive drugs at standard maintenance doses).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elsubrutinib Placebo/Upadacitinib Placebo | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) | Elsubrutinib Placebo/Upadacitinib 30 mg
Number analyzed (Participants) | 75 | 68 | 62
percentage of participants | 13.3 [5.6 to 21.0] | 30.9 [19.9 to 41.9] | 45.2 [32.8 to 57.5]
Statistical Analysis 1: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.007, Cochran-Mantel-Haenszel; Response Rate Difference = 16.7, 95% CI 2-sided [4.5 to 28.9]
Statistical Analysis 2: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs Elsubrutinib Placebo/Upadacitinib 30 mg; Elsubrutinib placebo/upadacitinib 30 mg vs elsubrutinib placebo/upadacitinib placebo; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Response Rate Difference = 31.0, 95% CI 2-sided [18.1 to 44.0]
Statistical Analysis 3: Comparison: ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) vs Elsubrutinib Placebo/Upadacitinib 30 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.068, Cochran-Mantel-Haenszel; Response Rate Difference = -13.7, 95% CI 2-sided [-28.4 to 1.0]

5. Secondary Outcome: Change From Baseline in Daily Prednisone Dose at Week 24
Description: Participants' current use of steroid therapy was assessed at each study visit, and the amount of daily prednisone was documented.
Time Frame: From Baseline to Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug with available data; Mixed-Effect Model Repeat Measurement was used. When 50% of planned participants had completed Week 24 or withdrawn from the study, the ABBV-599 Low Dose and elsubrutinib 60 mg treatment groups were terminated as these groups did not meet projected efficacy. Per protocol, terminated groups were removed from the efficacy analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg
Arm/Group | Elsubrutinib Placebo/Upadacitinib Placebo | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) | Elsubrutinib Placebo/Upadacitinib 30 mg
Number analyzed (Participants) | 56 | 54 | 48
mg | -0.65 [-1.57 to 0.28] | -0.45 [-1.38 to 0.48] | -0.62 [-1.60 to 0.36]
Statistical Analysis 1: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg); ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs elsubrutinib placebo/upadacitinib placebo The Mixed-Effect Model Repeat Measurement model included fixed effects of Tx, visit and Tx-by-visit interaction, stratification factors (Baseline corticosteroid dose > 10 mg prednisone-equivalent (≤ 10 mg or >10 mg), screening SLEDAI-2K (<10 or ≥ 10), baseline interferon score (high/low/NA, baseline immunosuppressant (yes/no)), and continuous fixed covariates of measurements at Baseline; Test type: Superiority; p = 0.710, Mixed-effect model repeat measurement; LS Mean Difference = 0.20, 95% CI 2-sided [-0.84 to 1.23], Standard Error of Mean 0.527
Statistical Analysis 2: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs Elsubrutinib Placebo/Upadacitinib 30 mg; Elsubrutinib placebo/upadacitinib 30 mg vs elsubrutinib placebo/upadacitinib placebo The Mixed-Effect Model Repeat Measurement model included fixed effects of Tx, visit and Tx-by-visit interaction, stratification factors (Baseline corticosteroid dose > 10 mg prednisone-equivalent (≤ 10 mg or >10 mg), screening SLEDAI-2K (<10 or ≥ 10), baseline interferon score (high/low/NA, baseline immunosuppressant (yes/no)), and continuous fixed covariates of measurements at Baseline; Test type: Superiority; p = 0.963, Mixed-effect model repeat measurement; LS Mean Difference = 0.03, 95% CI 2-sided [-1.05 to 1.10], Standard Error of Mean 0.545
Statistical Analysis 3: Comparison: ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) vs Elsubrutinib Placebo/Upadacitinib 30 mg; ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs elsubrutinib placebo/upadacitinib 30 mg The Mixed-Effect Model Repeat Measurement model included fixed effects of Tx, visit and Tx-by-visit interaction, stratification factors (Baseline corticosteroid dose > 10 mg prednisone-equivalent (≤ 10 mg or >10 mg), screening SLEDAI-2K (<10 or ≥ 10), baseline interferon score (high/low/NA, baseline immunosuppressant (yes/no)), and continuous fixed covariates of measurements at Baseline; Test type: Superiority; p = 0.754, Mixed-effect model repeat measurement; LS Mean Difference = 0.17, 95% CI 2-sided [-0.90 to 1.25], Standard Error of Mean 0.547

6. Secondary Outcome: Number of Flares Per Patient-year by Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA) SLEDAI Flare Index Through Week 24
Description: The SELENA SLEDAI flare index defines mild/moderate or severe SLE flares using the SLEDAI score, definitions of worsening signs and symptoms, treatment changes, and Physician's Global Assessment of Disease Activity.
Time Frame: From Baseline to Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug with available data; data as observed. When 50% of planned participants had completed Week 24 or withdrawn from the study, the ABBV-599 Low Dose and elsubrutinib 60 mg treatment groups were terminated as these groups did not meet projected efficacy. Per protocol, terminated groups were removed from the efficacy analyses.
Measure: Number (95% Confidence Interval); unit: Events per patient-year
Arm/Group | Elsubrutinib Placebo/Upadacitinib Placebo | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) | Elsubrutinib Placebo/Upadacitinib 30 mg
Number analyzed (Participants) | 75 | 68 | 62
Events per patient-year
  Mild/Moderate | 2.45 [1.92 to 2.99] | 1.39 [0.97 to 1.81] | 1.76 [1.28 to 2.25]
  Severe | 0.36 [0.16 to 0.56] | 0.26 [0.08 to 0.44] | 0.10 [-0.01 to 0.22]
  Overall | 2.81 [2.24 to 3.38] | 1.65 [1.20 to 2.10] | 1.87 [1.37 to 2.36]
Statistical Analysis 1: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg); Mild/Moderate ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs Elsubrutinib placebo/upadacitinib placebo A negative binomial regression model was used to assess treatment effect with treatment, visit, and stratification factors as covariates; Test type: Superiority; p = 0.002, Binomial regression; Rate difference = -1.06, 95% CI 2-sided [-1.74 to -0.39]
Statistical Analysis 2: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs Elsubrutinib Placebo/Upadacitinib 30 mg; Mild/Moderate Elsubrutinib placebo/upadacitinib 30 mg vs elsubrutinib placebo/upadacitinib placebo A negative binomial regression model was used to assess treatment effect with treatment, visit, and stratification factors as covariates; Test type: Superiority; p = 0.059, Binomial regression; Rate Difference = -0.69, 95% CI 2-sided [-1.41 to 0.03]
Statistical Analysis 3: Comparison: ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) vs Elsubrutinib Placebo/Upadacitinib 30 mg; Mild/Moderate ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs elsubrutinib placebo/upadacitinib 30 mg A negative binomial regression model was used to assess treatment effect with treatment, visit, and stratification factors as covariates; Test type: Superiority; p = 0.252, Binomial regression; Rate Difference = -0.37, 95% CI 2-sided [-1.01 to 0.27]
Statistical Analysis 4: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg); Severe ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs elsubrutinib placebo/upadacitinib placebo A negative binomial regression model was used to assess treatment effect with treatment, visit, and stratification factors as covariates; Test type: Superiority; p = 0.467, Binomial regression; Rate Difference = -0.10, 95% CI 2-sided [-0.37 to 0.17]
Statistical Analysis 5: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs Elsubrutinib Placebo/Upadacitinib 30 mg; Severe Elsubrutinib placebo/upadacitinib 30 mg vs elsubrutinib placebo/upadacitinib placebo A negative binomial regression model was used to assess treatment effect with treatment, visit, and stratification factors as covariates; Test type: Superiority; p = 0.033, Binomial regression; Rate Difference = -0.26, 95% CI 2-sided [-0.49 to -0.02]
Statistical Analysis 6: Comparison: ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) vs Elsubrutinib Placebo/Upadacitinib 30 mg; Severe ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs elsubrutinib placebo/upadacitinib 30 mg A negative binomial regression model was used to assess treatment effect with treatment, visit, and stratification factors as covariates; Test type: Superiority; p = 0.156, Binomial regression; Rate Difference = 0.15, 95% CI 2-sided [-0.06 to 0.37]
Statistical Analysis 7: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg); Overall ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs elsubrutinib placebo/upadacitinib placebo A negative binomial regression model was used to assess treatment effect with treatment, visit, and stratification factors as covariates; Test type: Superiority; p = 0.002, Binomial regression; Rate Difference = -1.16, 95% CI 2-sided [-1.89 to -0.44]
Statistical Analysis 8: Comparison: Elsubrutinib Placebo/Upadacitinib Placebo vs Elsubrutinib Placebo/Upadacitinib 30 mg; Overall Elsubrutinib placebo/upadacitinib 30 mg vs elsubrutinib placebo/upadacitinib placebo A negative binomial regression model was used to assess treatment effect with treatment, visit, and stratification factors as covariates; Test type: Superiority; p = 0.014, Binomial regression; Rate Difference = -0.95, 95% CI 2-sided [-1.70 to -0.19]
Statistical Analysis 9: Comparison: ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) vs Elsubrutinib Placebo/Upadacitinib 30 mg; Overall ABBV-599 High Dose (Elsubrutinib 60 mg/upadacitinib 30 mg) vs elsubrutinib placebo/upadacitinib 30 mg A negative binomial regression model was used to assess treatment effect with treatment, visit, and stratification factors as covariates; Test type: Superiority; p = 0.526, Binomial regression; Rate Difference = -0.22, 95% CI 2-sided [-0.89 to 0.46]

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; median time on follow-up was 337.0 days, 337.0 days, 338.5 days, 281.0 days, and 295.0 days for the placebo, ABBV-599 High Dose, upadacitinib, ABBV-599 Low Dose, and elsubrutinib groups, respectively.
Description: TEAEs and SAEs were collected from first dose of study drug until 30 days after last dose of study drug; mean time on treatment was 286.1 days, 289.8 days, 297.7 days, 226.4 days, and 228.6 days, for the placebo, ABBV-599 High Dose, upadacitinib, ABBV-599 Low Dose, and elsubrutinib groups, respectively.
Arm/Group | Elsubrutinib Placebo/Upadacitinib Placebo | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) | Elsubrutinib Placebo/Upadacitinib 30 mg | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) | Elsubrutinib 60 mg/Upadacitinib Placebo
All-Cause Mortality (participants affected / at risk) | 0/75 | 2/68 | 0/62 | 0/69 | 2/67
Serious Adverse Events (participants affected / at risk) | 13/75 | 7/68 | 13/62 | 9/69 | 7/67
Other Adverse Events (participants affected / at risk) | 39/75 | 38/68 | 35/62 | 28/69 | 36/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elsubrutinib Placebo/Upadacitinib Placebo (N=75) | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) (N=68) | Elsubrutinib Placebo/Upadacitinib 30 mg (N=62) | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) (N=69) | Elsubrutinib 60 mg/Upadacitinib Placebo (N=67)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
STRESS CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACCIDENTAL DEATH (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DISSEMINATED VARICELLA ZOSTER VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENDOCARDITIS BACTERIAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ESCHERICHIA SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENINGITIS TUBERCULOUS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MYCOPLASMA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PELVIC ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMOCYSTIS JIROVECII PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
PNEUMONIA FUNGAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS DISEASE ACTIVITY INDEX INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYSTEMIC LUPUS ERYTHEMATOSUS (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (2)
CENTRAL NERVOUS SYSTEM LUPUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RUPTURED CEREBRAL ANEURYSM (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BIPOLAR DISORDER (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUPUS NEPHRITIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BREAST MASS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSIVE URGENCY (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Clotted peripheral IV catheter in participant's arm
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elsubrutinib Placebo/Upadacitinib Placebo (N=75) | ABBV-599 High Dose (Elsubrutinib 60 mg/Upadacitinib 30 mg) (N=68) | Elsubrutinib Placebo/Upadacitinib 30 mg (N=62) | ABBV-599 Low Dose (Elsubrutinib 60 mg/Upadacitinib 15 mg) (N=69) | Elsubrutinib 60 mg/Upadacitinib Placebo (N=67)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 1 (1) | 1 (1) | 4 (4) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 6 (6) | 3 (4) | 4 (5) | 3 (4) | 2 (3)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
NAUSEA (Gastrointestinal disorders) | 6 (11) | 4 (4) | 4 (4) | 2 (2) | 6 (6)
VOMITING (Gastrointestinal disorders) | 3 (3) | 2 (3) | 4 (6) | 2 (2) | 2 (2)
FATIGUE (General disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 3 (3)
PYREXIA (General disorders) | 6 (6) | 3 (3) | 3 (3) | 2 (2) | 1 (1)
BRONCHITIS (Infections and infestations) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 8 (8) | 3 (3) | 7 (7) | 2 (2) | 8 (8)
HERPES ZOSTER (Infections and infestations) | 3 (3) | 7 (7) | 3 (3) | 3 (3) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 3 (3) | 6 (6) | 1 (1) | 5 (6) | 0 (0)
ORAL HERPES (Infections and infestations) | 1 (1) | 5 (11) | 3 (4) | 3 (3) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8 (10) | 7 (13) | 5 (6) | 5 (5) | 5 (6)
URINARY TRACT INFECTION (Infections and infestations) | 9 (10) | 8 (14) | 11 (15) | 5 (9) | 4 (4)
WEIGHT INCREASED (Investigations) | 1 (1) | 4 (8) | 1 (2) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 1 (1) | 2 (3) | 5 (5)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (3) | 1 (1) | 2 (2) | 2 (2)
HEADACHE (Nervous system disorders) | 9 (13) | 4 (4) | 2 (2) | 7 (8) | 10 (12)
INSOMNIA (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (4) | 2 (2) | 4 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-10-25): https://cdn.clinicaltrials.gov/large-docs/20/NCT03978520/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT03978520/SAP_001.pdf